CLINICAL TRIAL: NCT00039520
Title: A Phase II Trial Of Exisulind With Docetaxel In Patients With Metastatic Adenocarcinoma Of The Breast
Brief Title: Sulindac and Docetaxel in Treating Women With Metastatic or Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069390; P30CA006927 (NIH); FCCC-01031; FCCC-63723; NCI-G02-2080
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Sulindac

INTERVENTIONS:
Drug: docetaxel
Drug: sulindac

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining sulindac with docetaxel in treating women who have metastatic or recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of women with metastatic or recurrent adenocarcinoma of the breast treated with sulindac and docetaxel.
* Determine the time to progression of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive oral sulindac twice daily. Patients also receive docetaxel IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed within 3-4 weeks.

PROJECTED ACCRUAL: Approximately 12-33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Metastatic or recurrent disease
* Measurable disease

  * Bone only disease is not eligible
* No hematologic malignancy
* No carcinomatous meningitis and/or untreated or uncontrolled brain parenchymal disease

  * At least 8 weeks since prior therapy for brain parenchymal disease and patient must be asymptomatic from CNS disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Premenopausal or postmenopausal

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* One of the following:

  * SGOT and SGPT no greater than 2.5 times ULN AND
  * Alkaline phosphatase no greater than ULN OR
  * SGOT and SGPT no greater than ULN AND
  * Alkaline phosphatase no greater than 4 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No unstable angina
* No uncontrolled atrial or ventricular arrhythmias
* No congestive heart failure
* No uncontrolled hypertension

Other:

* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or contralateral breast cancer
* No active unresolved infection
* No poorly controlled diabetes mellitus
* No prior hypersensitivity reactions to sulindac or Polysorbate 80
* No peripheral neuropathy grade 2 or greater
* No active peptic ulcer disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent biological response modifiers
* No concurrent trastuzumab (Herceptin)

Chemotherapy:

* No more than 1 prior chemotherapy regimen in the adjuvant setting
* No more than 1 prior chemotherapy regimen for recurrent or metastatic disease
* No prior docetaxel
* Prior paclitaxel allowed
* At least 1 week since prior chronic sulindac
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent sulindac
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 1 week since prior antibiotics
* At least 4 weeks since prior investigational agents
* No other concurrent investigational drugs
* No other concurrent antineoplastic therapy
* No concurrent chronic (full dose for more than 2 weeks) nonsteroidal anti-inflammatory drugs (except ibuprofen or naproxen sodium), including cyclo-oxygenase-2 inhibitors and salicylates (e.g., aspirin, mesalamine, azodisalicylate, salsalate, or sulfasalazine)
* No concurrent parenteral antibiotics
* Concurrent low-dose aspirin for cardiovascular prevention allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-01; Primary Completion 2004-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Cianfrocca, DO, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States